CLINICAL TRIAL: NCT05115942
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Entecavir-based, Phase III Clinical Trial of Hydronidone Capsule in the Treatment of Liver Fibrosis Associated with Chronic Hepatitis B
Brief Title: Hydronidone for the Treatment of Liver Fibrosis Associated with Chronic Viral Hepatitis B Phase 3 Trial.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KDN-F351-202101
Record Dates: First submitted 2021-10-09; First posted 2021-11-10 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-08

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — hydronidone; 5-methyl-1-(4-hydroxylphenyl)-2-(1H)-pyridone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydronidone group (Experimental): Patients were orally received hydronidone capsules,3 capsules each time, t.i.d. for 52 weeks.
  Interventions: Drug: Hydronidone capsules
- The placebo group (Placebo Comparator): Patients were orally received placebo capsules,3 capsules each time, t.i.d. for 52 weeks.
  Interventions: Drug: The placebo capsules

INTERVENTIONS:
Drug: Hydronidone capsules — After randomization, the experimental group were orally received hydronidone capsules at a daily dose of 270 mg, 3 capsules each time, t.i.d,30 min before meals for 52 weeks.
  Other Names: F351
  Arms: Hydronidone group
Drug: The placebo capsules — After randomization, The control group were orally received placebo capsules at a daily dose of 270 mg, 3 capsules each time, t.i.d, 30 min before meals for 52 weeks.
  Other Names: N
  Arms: The placebo group

SUMMARY:
This study was a randomized, double-blind, placebo-controlled, entecavir basic treatment, multicentre clinical study.

The main objective of this study was to confirm the efficacy and safety of hydronidone in the treatment of chronic hepatitis B liver fibrosis.

DETAILED DESCRIPTION:
248 patients with chronic viral hepatitis B liver fibrosis were enrolled in this 52-week study, and randomized into hydronidone or placebo group. Each group has 124 patients. Both groups were treated with entecavir antiviral basic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years old (including 18 and 65 years old, based on the time of signing the written informed consent); gender is not limited.
2. History of chronic hepatitis B and/or hepatitis B surface antigen (HBsAg) positive≥6 months.
3. Percutaneous liver biopsy confirmed liver fibrosis (Ishak score ≥3).
4. Positive HBV DNA.
5. ALT < 8 x ULN (standard upper limit).
6. No antiviral therapy with interferon and/or nucleoside analogues within 3 months prior to enrollment.
7. 3 months before inclusion, he/she had not received any of the following proprietary Chinese medicines that may have anti-fibrosis effects: Fuzheng Huayu Capsule (tablet), Anluo Huayu Pill, compound Bijiaruangan tablet, etc.
8. The subject (or his/her sexual partner) had no pregnancy plan during the trial period and within 6 months after the trial, voluntarily used effective physical contraception, and had no sperm or egg donation plan.
9. Before the trial, they have understood the nature, significance, potential benefits, inconvenience and potential dangers of the trial in detail, and have voluntarily participated in the clinical trial, have good communication with the researchers, comply with the requirements of the whole study, and have signed a written informed consent form.

Exclusion Criteria:

1. Massive upper gastrointestinal hemorrhage within 3 months before enrolment.
2. Total bilirubin (TBiL) > 3×ULN, or 3×ULN < ALT < 8×ULN and TBiL > 2×ULN.
3. AFP > 100 μg/L although there was no indication of liver cancer.
4. Platelets (PLT) ≤60×109/L.
5. Prothrombin activity (PTA) < 50% or INR > 1.5.
6. Imaging showed obvious space-occupying lesions in the liver, suggesting tumor.
7. Body mass index (BMI) > 30 kg/m2.
8. Patients with decompensated liver cirrhosis and liver malignant tumor.
9. Patients with chronic hepatitis C or non-viral (alcoholic, non-alcoholic, drug, etc.) chronic hepatitis.
10. Serious diseases of cardiovascular, pulmonary, renal, endocrine, neurological and haematological systems, as well as mental disorders .
11. Women who are pregnant and/or breastfeeding.
12. Have participated in clinical trials of other drugs in the last 3 months.
13. The Investigator considers that there are any conditions that may affect the subjects' informed consent or adherence to the study protocol, or participation in the study may affect the study results or their own safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Ishak stage score of liver fibrosis by greater than or equal to 1 point after 52 weeks of treatment relative to baseline. | 52 weeks
  Clinically, the liver pathology scoring system, Ishak system, is widely used make a detailed and accurate assessment of the degree of parenchymal fibrosis or cirrhosis of the nontumorous liver. Ishak system uses a scale of 7 stages (scores 0-6) for the degree of fibrosis; the higher the score, the higher degree the severity of the disease.

SECONDARY OUTCOMES:
Change in liver inflammation grade by greater than or equal to 1 grade after 52 weeks of treatment relative to baseline but with no progression of fibrosis. | 52 weeks
  Scheuer score system is a liver pathology scoring system used for the diagnosis of liver inflammation and fibrosis pathology clinically; In the present trial, Scheuer system for scoring necroinflammatory activitt in chronic hepatitis will be used(G0-G4),the higher the score, the higher degree the severity of the disease.
Change in liver tissue inflammation grade by greater than or equal to 1 grade after 52 weeks of treatment relative to baseline. | 52 weeks
  Scheuer score system is a liver pathology scoring system used for the diagnosis of liver inflammation and fibrosis pathology clinically; In the present trial, Scheuer system for scoring necroinflammatory activitt in chronic hepatitis will be used(G0-G4),the higher the score, the higher degree the severity of the disease.
Change in liver stiffness measurement values via transient elastography LSM (kPa) | Screening period/baseline and weeks 12, 24, 36, and 52 after treatment .
  Change in liver stiffness measurement values via transient elastography LSM (kPa) values relative to baseline after 52 weeks of treatment.
Negative conversion (below the lower limit of detection) and the extent of decrease in HBV DNA | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Negative conversion (below the lower limit of detection) and the extent of decrease in HBV DNA after 52 weeks of treatment.
Normalization and the degree of improvement of the indicators of liver function ALT after 52 weeks of treatment. | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  ALT is one of the indicators to assess liver function and detect liver damage. When hepatic cells are affected by injury or disease, ALT is released into the blood, resulting in elevated ALT levels in the blood.
Safety endpoints:Laboratory examination（AFP test） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  AFP test: the serum AFP will be detected.
Safety endpoints:AE | 52 weeks
  Adverse events (AEs) refer to any adverse medical events that occur after the patient takes the study drug and can manifest as signs and symptoms, disease, or abnormal laboratory tests, but are not necessarily consequently related to the study drug.
  Information on AEs and Concomitant medications occurring in patients will be collected at the time points specified in the study schedule. AEs will be evaluated with reference to the Common Adverse Events Evaluation Criteria (NCI-CTCAE version 5.0).
Safety endpoints:Laboratory examination（Metabolic panel-AST） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Metabolic panel: The panel includes aspartate aminotransferase (AST)，which is one of the indicators to assess liver function and detect liver damage.
Safety endpoints:Laboratory examination（Metabolic panel-GGT） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Metabolic panel: The panel includes gamma-glutamyl transpeptidase (GGT),which is one of the indicators to assess liver function .
Safety endpoints:Laboratory examination（Metabolic panel-ALP） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Metabolic panel: The panel includes alkaline phosphatase (ALP),which is one of the indicators to assess liver function .
Safety endpoints:Laboratory examination（Metabolic panel-TP） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Metabolic panel: The panel includes total protein (TP), which is one of the indicators to assess liver function .
Safety endpoints:Laboratory examination（Metabolic panel-A） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Metabolic panel: The panel includes albumin (A) , which is one of the indicators to assess liver function .
Safety endpoints:Laboratory examination（Metabolic panel-TBiL） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Metabolic panel: The panel includes total bilirubin (TBiL) , which is one of the indicators to assess liver function .
Safety endpoints:Laboratory examination（Metabolic panel-DBiL） | Screening period/baseline and weeks 4, 8, 12, 24, 36, and 52 after treatment.
  Metabolic panel: The panel includes direct bilirubin (DBiL) , which is one of the indicators to assess liver function .

CONTACTS AND LOCATIONS:
Overall Officials: Lungen Lu, Dr., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Jun Cheng, Dr., Principal Investigator — Beijing Ditan Hospital
Locations (44):
- China (44):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing You 'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Tsinghua Changgeng Hospital, Beijing, Beijing, Beijing Municipality
  - Chongqing Public Health Medical Treatment Center (Chongqing Infectious Disease Hospital), Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fujian, Fujian
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - Lanzhou university first hospital, Lanzhou, Gansu
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong
  - Guizhou Provincial People's Hospital, Guizhou, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hangzhou Xixi Hospital (Hangzhou Sixth People's Hospital), Hangzhou, Hangzhou
  - The First Hospital of Hebei Medical University, Hebei, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Henan, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Zhengzhou Sixth People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Yueyang, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of SuZhou University, Suzhou, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Wuxi Fifth People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Zhenjiang Third People's Hospita, Zhenjiang, Jiangsu
  - Nanchang Ninth Hospital (Nanchang Central Hospital), Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Jilin, Jilin
  - Second Hospital of Jilin University, Jilin, Jilin
  - Yanbian University Affiliated Hospital, Yanbian, Jilin
  - Shanghai General Hospital,Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University Affiliated Tongren Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Traditional Chinese Medicine of Southwest Medical University, Luzhou, Sichuan
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No